CLINICAL TRIAL: NCT01635439
Title: Induction of Labour: A Comparison Between Propess Vaginal Delivery System and Prostin E2 Vaginal Suppositories, A Randomized Controlled Trial.
Brief Title: Prostin and Propess in Induction of Labor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: North West Armed Forces Hospital (Unknown)
Responsible Party: Principal Investigator, Mohamed Ellaithy, Lecturer of Obstetrics & Gynecology/ Consultant of Obstetrics & Gynecology AFHSR, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NWAFH2010-1
Record Dates: First submitted 2012-07-04; First posted 2012-07-09 (Estimated); Results first posted 2012-10-04 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-01

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Dinoprostone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propess (Active Comparator): Propess insert is a preparation of PGE2 packaged in a hydrogel polymer matrix and designed for slow intravaginal release of 10 mg dinoprostone at a rate of 0.3 mg/h.
  Interventions: Drug: Propess
- Prostin E2 (Active Comparator): PROSTIN E2 Vaginal Suppository, an oxytocic, contains dinoprostone as the naturally occurring prostaglandin E2 (PGE2)3 mg/suppository.
  Interventions: Drug: Prostin E2

INTERVENTIONS:
Drug: Propess — The vaginal insert is removed 24 h after the application. It is only to be removed earlier in case of the onset of active labour, the rupture of the membranes, or at the occurrence of hyperstimulation.
  Other Names: Intravaginal PGE2 insert
  Arms: Propess
Drug: Prostin E2 — 3 mg tab is placed in the posterior vaginal fornix. dose can be repeated every 6 hours till onset of active labour, the rupture of the membranes, or the occurrence of hyper-stimulation.
  Other Names: Dinoprostone (PGE2)vaginal tablets.
  Arms: Prostin E2

SUMMARY:
The purpose of the study was to compare the safety and efficacy of two agents used in induction of labor Propess (Controlled release dinoprostone, PGE2, pessary) and Prostin E2 (Dinoprostone vaginal Tablet).

DETAILED DESCRIPTION:
A controlled release hydrophilic matrix (Controlled Therapeutics Ltd., East Kilbride, Scotland) which provides a gradual release of dinoprostone (prostaglandin E2) was introduced in 1995 (Propess, Ferring Pharmaceuticals). This preparation is used for the initiation or enhancement of cervical ripening in women at or after term with a singleton pregnancy and a cephalic presentation. Prostaglandin E2 causes softening and dilatation of the cervix and subsequently produces uterine contractions which may induce labour.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 37 weeks or more
* Singleton pregnancy
* Cephalic presentation.

Exclusion Criteria:

* Previous cesarean section
* Any contraindication for vaginal delivery
* Suspected Cephalo-Pelvic Disproportion
* Unexplained antepartum Hemorrhage

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2010-12; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdelaziz, M.D., Principal Investigator — North West Armed Forces Hospital
Locations (1):
- NWAFH, North west Armed Forces Hospital, Tabuk, Tabuk Region, Saudi Arabia

REFERENCES:
- [Derived] Abdelaziz A, Mahmoud AA, Ellaithy MI, Abees SH. Pre-induction cervical ripening using two different dinoprostone vaginal preparations: A randomized clinical trial of tablets and slow release retrievable insert. Taiwan J Obstet Gynecol. 2018 Aug;57(4):560-566. doi: 10.1016/j.tjog.2018.06.016. PMID 30122579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 290 women were assessed for eligibility, 62 women were excluded (35 did not meet the inclusion criteria, 21 declined to participate and 6 refused induction of labor as a method of delivery)
Pre-assignment Details: Among the 228 women who met the eligibility criteria, 7 went into spontaneous labor and 4 had pathological Cardiotocography (CTG), so were excluded from being assigned to one of the treatment groups. After allocation 17 women were excluded from the analysis (15 refused to continue the induction of labor and had 5 incomplete records).
Groups:
- Propess: Propess insert is a preparation of PGE2 packaged in a hydrogel polymer matrix and designed for slow intravaginal release of 10 mg dinoprostone at a rate of 0.3 mg/h over 12 h.
Period: Overall Study
Arm/Group | Propess | Prostin E2
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propess | Prostin E2 | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (4.3) | 26.8 (5.1) | 26.4 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 200
  Male | 0 | 0 | 0
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 23 (2.7) | 23.5 (3.5) | 23.3 (3.1)
Parity [Number; unit: participants] — Parity is the number times a woman has given birth to a fetus with a gestational age of 24 weeks or more, regardless of whether the child was born alive or was stillborn. (e.g., P3 is 3 births), a multiple birth considered as a single parous experience
  participants
    P0 | 44 | 49 | 93
    P1 | 20 | 23 | 43
    P2 | 20 | 14 | 34
    P3 | 11 | 8 | 19
    P4 | 3 | 3 | 6
    P5 | 2 | 3 | 5
Gestational age [Mean (Standard Deviation); unit: weeks] — For the purpose of pregnancy dating, Gestational age refers to the pregnancy duration in weeks calculated from the date of the last menstrual period.
  weeks | 40.6 (0.9) | 40.4 (1.3) | 40.5 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Induction to Delivery Interval
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Propess | Prostin E2
Number analyzed (Participants) | 100 | 100
hours | 22.3 (5.7) | 21.2 (5.3)

2. Secondary Outcome: Induction to Onset of Labor Interval
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Propess | Prostin E2
Number analyzed (Participants) | 100 | 100
hours | 18.8 (5.3) | 17.7 (5.4)

3. Secondary Outcome: Uterine Hyper-stimulation Rate
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Propess | Prostin E2
Number analyzed (Participants) | 100 | 100
participants | 1 | 1

4. Secondary Outcome: Need for Syntocinon Augmentation
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Propess | Prostin E2
Number analyzed (Participants) | 100 | 100
participants | 5 | 10

5. Secondary Outcome: Normal Vaginal Delivery Rate
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Propess | Prostin E2
Number analyzed (Participants) | 100 | 100
participants | 79 | 85

ADVERSE EVENTS:
Arm/Group | Propess | Prostin E2
Serious Adverse Events (participants affected / at risk) | 1/100 | 2/100
Other Adverse Events (participants affected / at risk) | 14/100 | 13/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propess (N=100) | Prostin E2 (N=100)
Cord pH < 7.1 (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propess (N=100) | Prostin E2 (N=100)
Maternal adverse outcomes (Pregnancy, puerperium and perinatal conditions) | 12 (12) | 13 (13)
Apgar score < 7 (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Uterine tachysystole (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No